CLINICAL TRIAL: NCT02892812
Title: A Single-blind, Single-center, Randomized, Active-controlled, Parallel Group, Phase I Study to Evaluate the Safety and Immunogenicity of Intramuscular Single Injection With LBVE013 (Pneumococcal 13-valent Conjugate Vaccine [Diphtheria CRM197 Protein]), LBVE014 (Pneumococcal 14-valent Conjugate Vaccine [Diphtheria CRM197 Protein]) or Prevnar13 in Healthy Adults
Brief Title: A Phase I Clinical Trial of a 13-valent Pneumococcal Conjugate Vaccine and 14-valent Pneumococcal Conjugate Vaccine in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LG-VECL001
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- LBVE013 (Experimental): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine
- LBVE014 (Experimental): 14-valent pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine
- Prevnar13 (Active Comparator): 13-valent pneumococcal conjugate vaccine
  Interventions: Biological: Pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: Pneumococcal conjugate vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of LBVE013 (Pneumococcal 13-valent conjugate vaccine [diphtheria CRM197 protein]) or LBVE014 (Pneumococcal 14-valent conjugate vaccine [diphtheria CRM197 protein]) in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult older than 19 years old and younger than 50 years old
* A subject who was informed of the purpose, method, and efficacy of the clinical study and signed the written informed consent form

Exclusion Criteria:

* A subject who participated in other clinical studies within 3 months before screening
* A subject who was vaccinated with other vaccines within 4 weeks before screening, or who is expected to receive other vaccination during the clinical study period
* A subject with medical history of hypersensitive reactions (e.g. anaphylaxis) to the test drug or its ingredients
* A subject who received immunoglobulin or blood-derived materials within 3 months before screening
* A subject with immunologic function disorders including congenital or acquired immunodeficiency disorders
* A subject who is receiving immunosuppressive therapy or drugs that can affect immunological reaction
* A subject with pyrexia of over 38 Celsius degrees on the day of the vaccination with the investigational products
* A subject with medical history of Invasive Pneumococcal Disease (IPD) or pneumonia caused by Streptococcus pneumoniae
* A subject who was vaccinated with any pneumococcal vaccine before screening
* A subject who received the vaccine containing diphtheria toxoid within 6 months before screening (e.g. adult Td vaccine)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events | Baseline(pre-vaccination) up to 7 days after vaccination
Unsolicited adverse events | Baseline(pre-vaccination) up to 4 weeks after vaccination
Immediate reactions after vaccination | Baseline(pre-vaccination) up to 30 minutes after vaccination

SECONDARY OUTCOMES:
Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 4 weeks After Vaccination | 4 weeks after vaccination
Proportion of subjects achieving 4-fold rise in Pneumococcal Opsonophagocytic Activity (OPA) titer at 4 weeks after vaccination | 4 weeks after vaccination
Serotype-Specific Pneumococcal IgG antibody Geometric Mean Concentrations (GMCs) 4 weeks After Vaccination | 4 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided